CLINICAL TRIAL: NCT03746067
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Effects of Food on the Absorption of TS-134 Administered Orally to Healthy Male and Female Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Doses of TS-134 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical R&D Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TS134-US101
Record Dates: First submitted 2018-10-18; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
Keywords: TS-134, CSF

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TS-134 (Experimental): Healthy adult subjects will be prospectively assigned to 1 of 4 cohorts. Within each cohort, 8 subjects will be randomized in a 3:1 ratio (6 active + 2 placebo) per cohort to receive TS-134 or placebo as a single oral dose solution. All cohorts will be dosed in a fasted state except for the 2nd and 4th (food effect) cohorts, which will be dosed first in a fasted state, and then in a fed state, in a single crossover design conducted with a washout between two periods. In the 3rd (CSF) cohort, 8 subjects will receive one dose level of TS-134 as a single-blind dosing assignment; there will be no placebo dosing.
  Interventions: Drug: TS-134
- Placebo (Placebo Comparator): Healthy adult subjects will be prospectively assigned to 1 of 4 cohorts. Within each cohort, 8 subjects will be randomized in a 3:1 ratio (6 active + 2 placebo) per cohort to receive TS-134 or placebo as a single oral dose solution. All cohorts will be dosed in a fasted state except for the 2nd and 4th (food effect) cohorts, which will be dosed first in a fasted state, and then in a fed state, in a single crossover design conducted with a washout between two periods. In the 3rd (CSF) cohort, the 8 subjects will receive one dose level of TS-134 as a single-blind dosing assignment; there will be no placebo dosing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TS-134 — 5 mg, 10 mg, or 20 mg oral solution
  Arms: TS-134
Drug: Placebo — Matched Placebo oral solution
  Arms: Placebo

SUMMARY:
This is a Phase 1a study involving single oral dose of TS-134 in healthy male and female subjects. The safety, tolerability and pharmacokinetics of single dose of TS-134 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female participants between 18 and 55 years of age
* Body weight greater than or equal to 45 kg
* Body Mass Index (BMI) greater than or equal to 18 and less than or equal to 30 kg/m^2

Exclusion Criteria:

* Female participants who are pregnant, intend to become pregnant, or are breastfeeding
* Clinically significant abnormal physical examination, 12-lead electrocardiogram (ECG) OR cardiac telemetry prior to dosing.
* Significant history or presence of hepatic, renal, cardiovascular, pulmonary, gastrointestinal, hematological, locomotor, immunologic, ophthalmologic, metabolic or oncological disease.
* History or presence of psychiatric or neurologic disease or condition
* History of alcohol or drug abuse
* Any participant who currently uses or has used tobacco or tobacco-containing products for at least one month prior to screening
* Participated in strenuous exercise within 48 hours prior to study start (initial dosing) and/or are unwilling to avoid strenuous exercise at any time throughout the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2016-01-13 (Actual); Study Completion 2016-01-13 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events | Day 1 to Day 7
TS-134 Plasma Pharmacokinetic Profile - Cmax | Day 1: predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  Maximum plasma concentration
TS-134 Plasma Pharmacokinetic Profile - AUC(0-last) | Day 1: predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  Area under the concentration vs. time curve from time zero to last measurable concentration
TS-134 Plasma Pharmacokinetic Profile - tmax | Day 1: predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  Time to maximum plasma concentration
TS-134 Plasma Pharmacokinetic Profile - t1/2 | Day 1: predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  Apparent terminal elimination half-life
TS-134 Plasma Pharmacokinetic Profile - CL/F | Day 1: predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  Apparent clearance following oral administration
TS-134 Plasma Pharmacokinetic Profile - Vd/F | Day 1: predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  Apparent volumes of distribution following oral administration

SECONDARY OUTCOMES:
TS-134 Cerebral Spinal Fluid (CSF) Pharmacokinetic Profile - Cmax | Day 1: predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose
  Maximum CSF concentration
TS-134 CSF Pharmacokinetic Profile - AUC(0-last) | Day 1: predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose
  Area under the CSF concentration vs. time curve from time zero to last measurable concentration
TS-134 CSF Pharmacokinetic Profile - tmax | Day 1: predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose
  Time to maximum CSF concentration
TS-134 CSF Pharmacokinetic Profile - t1/2 | Day 1: predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose
  Apparent terminal elimination half-life (CSF)
TS-134 CSF Pharmacokinetic Profile - CL/F | Day 1: predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose
  Apparent clearance (CSF) following oral administration
TS-134 CSF Pharmacokinetic Profile - Vd/F | Day 1: predose, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 24 hours post-dose
  Apparent volumes of distribution (CSF) following oral administration

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical R&D Inc.
Locations (1):
- PAREXEL - Early Phase Clinical Unit-Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No